CLINICAL TRIAL: NCT06073756
Title: Neutrophil-lymphocyte and Platelet-lymphocyte Ratios and Their Relations to Vascular Comlications and Glycemic Control in Patients With Type 2 Diabetes Attending The Diabetes Center of Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ammar Ashraf fathy, Ammar Ashraf, Assiut University
Other Study IDs: NLR and PLR and in type 2 DM
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Vascular Complication, Diabetic
Keywords: Neutrophils to lymhocyte ratio and platelets to lymhocyte ratio
MeSH Terms: conditions — Diabetic Angiopathies | interventions — Albumins; Neural Conduction; Caves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Type 2 diabetes mellitus (T2DM) patients with good glycemic control and have HBA1C <7and ages ranging from ≥18 old.
  Interventions: Radiation: Echocardiogram
- 2: Type 2 diabetes mellitus (T2DM) patients with poor glycemic control and have HBA1C ≥7 and ages rang from ≥ 18 years old
  Interventions: Radiation: Echocardiogram

INTERVENTIONS:
Radiation: Echocardiogram — Evaluate PLR and NLR and their assiotation to vascular complications and glycemic control in type 2 DM
  Other Names: ALB / cr ratio; Fundus examination; ECG; Doppler on lower limbs; Nerve conduction; Echo

SUMMARY:
Evaluate PLR and NLR and their assiotation to vascular complications and glycemic control in type 2 DM

DETAILED DESCRIPTION:
Vascular complications of DM result from various disorders including metabolic, cellular, and blood disturbances. Excessive production of pro-inflammatory adipokines from adipose tissue, resulting in low-grade chronic inflammation, causing insulin resistance (IR) and type 2 DM [3]. Hematological changes affecting the red blood cells (RBCs), white blood cells (WBCs), platelet function, and the coagulation factors are detected to be associated with DM . It is important to add that, high WBC count, one of the chief components of inflammatory process, sharing to atheroscle-rosis development and cardiovascular diseases (CVD) . Lately, the neutrophil-to-lymphocyte (N/L) and the platelet-to-lymphocyte (P/L) ratios, were offered as markers of inflammation in cardiac diseases, neoplasms and diabetes-related complications . Moreover, high leucocyte counts have been used as diagnostic and prognostic markers in vascular complication of diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (T2DM) patients with good glycemic control and have HBA1C <7and ages ranging from ≥18 old. And poor glycemic control and have HBA1C ≥7 and ages rang from ≥ 18 years old

Exclusion Criteria:

* Patients with, type 1 diabetes mellitus

  1. Idiopathic thrombocytopenic purpura,
  2. liver cell failure
  3. Myeloproliferative neoplasm
  4. patients on anticoagulant drugs , anti platelet drugs or on steroids were excluded from the study

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Evaluate PLR and NLR and their assiotation to vascular complications and glycemic control in type 2 DM
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Neutrophil-to-lymphocyte ratio and platelets to lymphocytes ratio | Basline
  Measurement of Neutrophils to lymhocyte ratio and platelets to lymhocyte ratio in patients with type 2 DM

SECONDARY OUTCOMES:
HbA1c with good glycemic control and have HBA1C lower than 7and poor glycemic control and have HBA1C higher than 7with prescence or abscence of vascular complications | Basline
  Evaluate PLR and NLR and their assiotation to vascular complications and glycemic control in type 2 DM